CLINICAL TRIAL: NCT02233010
Title: Usefulness of Neutrophil Gelatinase-associated Lipocalin(NGAL) to Confirm Acute Kidney Function Decrease of the Patients Who Had Non-cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Hoseok Koo, Hoseok Koo, Inje University
Other Study IDs: postOPNGAL01
Record Dates: First submitted 2014-09-01; First posted 2014-09-08 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- kidney function normal group: kidney function normal group : defined by the normal level of NGAL after post operation 4hrs
  Interventions: Other: The level of NGAL after pre op,post op 4hr, post op 12hr
- kidney function decreased group: kidney function decreased group : defined by the increased level of NGAL after post operation 4hrs
  Interventions: Other: The level of NGAL after pre op,post op 4hr, post op 12hr

INTERVENTIONS:
Other: The level of NGAL after pre op,post op 4hr, post op 12hr

SUMMARY:
Although post-op renal function decrease is determined by serum creatinine, serum creatinine has disadvantages that it increases a long time after renal function decrease and it has various increasing time based on the level of renal function. Neutrophil Gelatinase-associated Lipocalin (NGAL's) usefulness as an evidence for acute kidney damage occurring from post-op cardiac surgery, being critical patients and contrast medium use is already proven.

But NGAL's usefulness for renal function after non-cardiac surgery is not proven and especially, NGAL's usefulness for renal injury after non-cardiac surgery in chronic renal disease patients is not proven.Therefore, the investigators will study about renal function decrease after non-cardiac surgery with NGAL and serum creatinine.

ELIGIBILITY:
Inclusion Criteria:

* 43 patients who had non-cardiac surgery in Seoul Paik Hospital.

Exclusion Criteria:

* have viral hepatitis and Aspartate aminotransferase, Alanine aminotransferase > 2 time of normal level
* severe lung disease
* severe heart failure ( Ejection Fraction < 40% )
* pregnancy

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 43 patients who had non-cardiac surgery in Seoul Paik Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
serum NGAL level | up to post operation 12 hours